CLINICAL TRIAL: NCT05421442
Title: A Nationwide Post-marketing Study on the Safety of Abatacept Treatment in Denmark Using the DANBIO Register
Brief Title: A Post-marketing Study on the Safety of Abatacept Treatment in Denmark Using the Danish Database
Acronym: DANBIO
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-803; EUPAS31532 (Registry Identifier: EU PAS Register)
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis (RA); Psoriatic Arthritis (PsA)
Keywords: Abatacept; Orencia; Malignancies; Long-term safety follow-up
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Abatacept Group: Participants with established rheumatoid arthritis (RA) or psoriatic arthritis (PsA) and receiving abatacept
- Non-targeted Disease Modifying Anti-rheumatic Drug (DMARD) Group: Participants with established RA or PsA and not previously treated with any targeted disease modifying anti-rheumatic drugs (DMARDs) and who start treatment with a non-targeted DMARD
- Targeted DMARD Group: Participants with established RA or PsA and previously treated without abatacept who start treatment with targeted DMARDs

SUMMARY:
The purpose of this study is to expand on the ongoing post-marketing monitoring of abatacept to include all participants with rheumatoid arthritis (RA) and psoriatic arthritis (PsA) treated with abatacept captured in Danish Database for Biologic Therapies (DANBIO).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis (RA) or psoriatic arthritis (PsA)
* Receiving treatment with abatacept
* Receiving treatment with non-targeted DMARD
* Receiving treatment with targeted DMARD

Exclusion Criteria:

-Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with RA or PsA who are enrolled in the Danish Database for Biologic Therapies (DANBIO) register in Denmark and were receiving abatacept, non-targeted DMARDs, or targeted DMARDs between January 2007 and December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 38396 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence Rates of Overall Malignancies | Up to 5 years
Incidence Rates of Melanoma | Up to 5 years
Incidence Rates of Non-melanoma Skin Cancer | Up to 5 years
Incidence Rates of Basal Cell Carcinoma | Up to 5 years
Incidence Rates of Squamous Cell Carcinoma | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Lawrenceville, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html